CLINICAL TRIAL: NCT04494126
Title: Effect of Perioperative Tranexamic Acid on Blood Loss During Management of Maxillofacial Trauma: A Randomized Double Blind Clinical Trial
Brief Title: Effect of Perioperative Tranexamic Acid on Blood Loss During Management of Maxillofacial Trauma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: College of Medical Sciences Teaching Hospital. Nepal (Other)
Responsible Party: Principal Investigator, Ashutosh Kumar Singh, Associate professor, College of Medical Sciences Teaching Hospital. Nepal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CMSNepal1
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Blood Loss
Keywords: Maxillofacial trauma; blood loss
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, Parallel assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the anaesthesiologist who is administering the medications is unmasked until completion of the data collection period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (Experimental): Experimental: TXA Group One gram of intravenous tranexamic acid (TXA) in normal saline (50cc) given over 15 minutes starting just prior to skin incision, and repeated 6 hours later in the postoperative period.
  Interventions: Drug: Tranexamic acid
- Placebo (Placebo Comparator): Placebo Comparator: Control Group Intravenous normal saline (50cc) given over 15 minutes starting just prior to skin incision, and repeated 6 hours later in the postoperative period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic acid — Drug: Tranexamic Acid Injectable Solution the drug will be given to patients intravenously at a dose of 10mg/kg pre-operatively after induction on general anesthesia before incision.
  Other Names: Injection TXA 1 gram
  Arms: Tranexamic acid
Drug: Placebo — Other: Placebo (normal saline 0.9%) An equivalent amount of normal saline (0.9%) will be given to the patient pre-operatively after induction of general anesthesia. The amount of saline given will correspond to the same amount of fluid which would have been given had the patient been in the intervention group.
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
This is a prospective, randomized, double-blind study investigating whether intravenous tranexamic acid has any effect on blood loss during maxillofacial trauma surgery, or the subsequent postoperative sequelae. Intraoperative bleeding and postoperative ecchymosis and edema are objectively rated and complications are noted.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind pilot study investigating whether intravenous tranexamic acid has any effect on blood loss during maxillofacial trauma surgery, or the subsequent postoperative sequelae. Intraoperative bleeding is calculated from anaesthesia chart and recorded in ml. Postoperative ecchymosis and bleeding are recorded as dichotomous events (yes/no) and are subjectively rated by both patient and surgeon on postoperative days 1and 2. Any surgical or postoperative complications are noted. Scores are aggregated for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ORIF under GA for Maxillofacial fractures
* Patients between with ages of 16-65
* No cardiac comorbidities (hypertension, congenital heart malformation)
* No known coagulopathy
* No regular prescription medication altering normal blood coagulation (NSAIDs, other anticoagulants)
* ASA I and II patients

Exclusion Criteria:

* Patients younger than 16 and older than 65
* Patients with known coagulopathy
* Patients with cardiac comorbidities
* Patients with a family history of bleeding disorders
* ASA III or higher

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-08-15 (Estimated); Primary Completion 2021-10-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss | Surgical period
  Measured and recorded from the anaesthesia patient chart

SECONDARY OUTCOMES:
Postoperative bleeding event | upto 48 hours after surgery
  postoperative bleeding and ecchymosis subjectively reported by patient and assessed by clinician, recorded as a dichotomous outcome.

OTHER OUTCOMES:
Complications if any during surgery and upto 48 hours after surgery | upto 48 hours after surgery
  complications related to surgery as reported by patient and clinician

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Yadav, MD, Study Director — College of Medical Sciences Teaching hospital, Bharatpur, Nepal

IPD SHARING:
Plan to Share IPD: No
The data will be used for internal use only. Any patient identifier will be removed from the final master chart before statistical analysis.